CLINICAL TRIAL: NCT02574481
Title: A Randomized Trial Comparing the ELUVIA™ Drug-eluting Stent Versus Zilver® PTX® Stent for Treatment of Superficial Femoral and/or Proximal Popliteal Arteries
Brief Title: ELUVIA™ Drug-eluting Stent Versus Zilver® PTX® Stent
Acronym: IMPERIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2063
Record Dates: First submitted 2015-09-22; First posted 2015-10-14 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Atherosclerosis of Native Arteries of the Extremities
Keywords: atherosclerosis; Superficial Femoral Artery (SFA); Proximal Popliteal Artery (PPA); lower extremities; stenting; paclitaxel
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ELUVIA Stent Implantation (Experimental): Percutaneous stent placement in the SFA/PPA
  Interventions: Device: ELUVIA (Stent Implantation)
- Zilver PTX Stent Implantation (Active Comparator): Percutaneous stent placement in the SFA/PPA
  Interventions: Device: Zilver PTX (Stent Implantation)

INTERVENTIONS:
Device: ELUVIA (Stent Implantation) — Drug-eluting self-expanding stent implantation during the index procedure.
  Arms: ELUVIA Stent Implantation
Device: Zilver PTX (Stent Implantation) — Drug-eluting self-expanding stent implantation during the index procedure.
  Arms: Zilver PTX Stent Implantation

SUMMARY:
The primary objective of this trial is to evaluate the safety and effectiveness of the Boston Scientific Corporation (BSC) ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions up to 140 mm in length.

Long Lesion Substudy: to evaluate the safety and effectiveness of the Boston Scientific Corporation (BSC) ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.

DETAILED DESCRIPTION:
Atherosclerosis is a systemic disease that has become increasingly recognized in the expanding elderly population as a significant cause of morbidity and mortality. Atherosclerosis in the vessels of the lower extremities can cause a variety of symptoms ranging from intermittent claudication to ischemic rest pain and critical ischemia with major tissue loss. Typically, femoropopliteal lesions have been difficult to successfully treat with endovascular therapy because the disease is often diffuse and located in an area of the body subject to significant mobility stresses such as extension, contraction, compression, elongation, flexion and torsion.

The IMPERIAL trial is a global, prospective, multi-center trial. Approximately 525-535 subjects will be enrolled at up to 75 study centers worldwide. Regions participating include the United States, Canada, European Union, Japan and New Zealand.

The trial consists of a prospective, multicenter, 2:1 randomized (ELUVIA vs Zilver PTX), controlled, single-blind, non-inferiority trial (RCT), a concurrent, non-blinded, non-randomized, single-arm, pharmacokinetic (PK) substudy and a concurrent, non-blinded, non-randomized, Long Lesion substudy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 and older.
2. Subject (or Legal Guardian if applicable) is willing and able to provide consent before any study-specific test or procedure is performed, signs the consent form, and agrees to attend all required follow-up visits. NOTE: For subjects less than 20 years of age enrolled at a Japanese center, the subject's legal representative, as well as the subject, must provide written informed consent.
3. Chronic, symptomatic lower limb ischemia defined as Rutherford categories 2, 3 or 4.
4. Stenotic, restenotic or occlusive lesion(s) located in the native SFA and/or PPA:

   * Degree of stenosis ≥ 70% by visual angiographic assessment
   * Vessel diameter ≥ 4 and ≤ 6 mm
   * Total lesion length (or series of lesions) ≥ 30 mm and ≤ 140 mm (Note: Lesion segment(s) must be fully covered with one ELUVIA stent or up to two Zilver PTX stents)
   * Long Lesion Substudy: Total lesion length (or series of lesions) >140 mm and ≤ 190 mm (Note: Lesion segment(s) will require overlapping of two ELUVIA stents).
   * For occlusive lesions requiring use of re-entry device, lesion length ≤ 120 mm
   * Long Lesion Substudy: For occlusive lesions requiring use of re-entry device, lesion length > 120 mm and ≤ 170 mm
   * Target lesion located at least three centimeters above the inferior edge of the femur
5. Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot with no planned intervention.

Exclusion Criteria:

1. Previously stented target lesion/vessel.
2. Target lesion/vessel previously treated with drug-coated balloon <12 months prior to randomization/enrollment.
3. Subjects who have undergone prior surgery of the SFA/PPA in the target limb to treat atherosclerotic disease.
4. Use of atherectomy, laser or other debulking devices in the target limb SFA/PPA during the index procedure.
5. History of major amputation in the target limb.
6. Documented life expectancy less than 24 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the clinical trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the clinical trial.
7. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
8. Known hypersensitivity/allergy to the investigational stent system or protocol related therapies (e.g., nitinol, paclitaxel, or structurally related compounds, polymer or individual components, and antiplatelet, anticoagulant, thrombolytic medications).
9. Platelet count <80,000 mm3 or >600,000 mm3 or history of bleeding diathesis.
10. Concomitant renal failure with a serum creatinine >2.0 mg/dL.
11. Receiving dialysis or immunosuppressant therapy.
12. History of myocardial infarction (MI) or stroke/cerebrovascular accident (CVA) within 6 months prior to randomization/enrollment.
13. Unstable angina pectoris at the time of randomization/enrollment.
14. Pregnant, breast feeding, or plan to become pregnant in the next 5 years.
15. Current participation in another investigational drug or device clinical study that has not completed the primary endpoint at the time of randomization/enrollment or that clinically interferes with the current study endpoints (Note: studies requiring extended follow-up for products that were investigational, but have become commercially available since then are not considered investigational studies).
16. Septicemia at the time of randomization/enrollment.
17. Presence of other hemodynamically significant outflow lesions in the target limb requiring intervention within 30 days of randomization/enrollment.
18. Presence of aneurysm in the target vessel.
19. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to randomization/enrollment.
20. Perforated vessel as evidenced by extravasation of contrast media prior to randomization/enrollment.
21. Heavily calcified lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Main Line Health; Stefan Müller-Hülsbeck, Prof, Principal Investigator — Ev. Luth. Diakonissenanstalt Flensburg
Locations (68):
- United States (42):
  - Yuma Regional Medical Center, Yuma, Arizona
  - University of California, Davis Medical Center, Sacramento, California
  - Florida Research Network, LLC, Gainesville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - MediQuest Research at Munroe Regional Medical Center, Ocala, Florida
  - Baptist Hospital, Pensacola, Florida
  - University Hospital, Augusta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Francis Medical Center, Peoria, Illinois
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Maine Medical Center, Portland, Maine
  - Steward St. Elizabeth's Medical Center of Boston, Inc., Boston, Massachusetts
  - Northern Michigan Hospital, Petoskey, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Alegent Creighton Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - New York University Medical Center, New York, New York
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - LakeWest Hospital/Northeast Ohio Vascular Associates, Inc., Willoughby, Ohio
  - Providence St. Vincents Medical Center, Portland, Oregon
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - University Surgical Associates, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - Texas Health Presbyterian Hospital, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Aspirus Heart and Vascular Institute - Research and Education, Wausau, Wisconsin
- Austria (3):
  - Medical University Graz, Department of Radiology, Graz
  - Allgemeines Krankenhaus AKH, Vienna
  - Hanusch Hospital, Vienna
- Belgium (3):
  - Ziekenhuis oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Fleurimont Hospital, Sherbrooke, Quebec
- Germany (5):
  - Universitäts-Herzzentrum Bad Krozingen, Bad Krozingen
  - Center for Diagnostic Radiology and Minimally Invasive Therapy at The Jewish Hospital Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Ev. Luth. Diakonissenanstalt Flensburg, Flensburg
  - Universität Leipzig, Leipzig
- Japan (10):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Takatsu General Hospital, Kawasaki, Kanagawa
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Toho University Ohashi Medical Center, Meguro City, Tokyo
  - The Jikei University Hospital, Minato, Tokyo
  - Fukuoka Sanno Hospital, Fukuoka
  - Morinomiya Hospital, Osaka
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Clinical Trials NZ, Hamilton

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Iida O, Fujihara M, Kawasaki D, Mori S, Yokoi H, Miyamoto A, Kichikawa K, Nakamura M, Ohki T, Diaz-Cartelle J, Muller-Hulsbeck S, Gray WA, Soga Y. 24-Month Efficacy and Safety Results from Japanese Patients in the IMPERIAL Randomized Study of the Eluvia Drug-Eluting Stent and the Zilver PTX Drug-Coated Stent. Cardiovasc Intervent Radiol. 2021 Sep;44(9):1367-1374. doi: 10.1007/s00270-021-02901-6. Epub 2021 Jul 7. PMID 34235560
- [Derived] Muller-Hulsbeck S, Benko A, Soga Y, Fujihara M, Iida O, Babaev A, O'Connor D, Zeller T, Dulas DD, Diaz-Cartelle J, Gray WA. Two-Year Efficacy and Safety Results from the IMPERIAL Randomized Study of the Eluvia Polymer-Coated Drug-Eluting Stent and the Zilver PTX Polymer-free Drug-Coated Stent. Cardiovasc Intervent Radiol. 2021 Mar;44(3):368-375. doi: 10.1007/s00270-020-02693-1. Epub 2020 Nov 22. PMID 33225377
- [Derived] Golzar J, Soga Y, Babaev A, Iida O, Kawasaki D, Bachinsky W, Park J, Prem JT, Vermassen F, Diaz-Cartelle J, Muller-Hulsbeck S, Gray WA. Effectiveness and Safety of a Paclitaxel-Eluting Stent for Superficial Femoral Artery Lesions up to 190 mm: One-Year Outcomes of the Single-Arm IMPERIAL Long Lesion Substudy of the Eluvia Drug-Eluting Stent. J Endovasc Ther. 2020 Apr;27(2):296-303. doi: 10.1177/1526602820901723. Epub 2020 Jan 28. PMID 31989856
- [Derived] Soga Y, Fujihara M, Iida O, Kawasaki D, Hirano K, Yokoi H, Miyamoto A, Kichikawa K, Nakamura M, Ohki T, Diaz-Cartelle J, Gray WA, Muller-Hulsbeck S. Japanese Patients Treated in the IMPERIAL Randomized Trial Comparing Eluvia and Zilver PTX Stents. Cardiovasc Intervent Radiol. 2020 Feb;43(2):215-222. doi: 10.1007/s00270-019-02355-x. Epub 2019 Nov 5. PMID 31690980
- [Derived] Gray WA, Keirse K, Soga Y, Benko A, Babaev A, Yokoi Y, Schroeder H, Prem JT, Holden A, Popma J, Jaff MR, Diaz-Cartelle J, Muller-Hulsbeck S; IMPERIAL investigators. A polymer-coated, paclitaxel-eluting stent (Eluvia) versus a polymer-free, paclitaxel-coated stent (Zilver PTX) for endovascular femoropopliteal intervention (IMPERIAL): a randomised, non-inferiority trial. Lancet. 2018 Oct 27;392(10157):1541-1551. doi: 10.1016/S0140-6736(18)32262-1. Epub 2018 Sep 24. PMID 30262332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 524 subjects have been enrolled in the IMPERIAL trial, including 465 subjects in the RCT, 50 subjects in the LL substudy and 13 subjects in the PK substudy. There were 4 subjects enrolled in both the PK and Long Lesion substudy.
Groups:
- Long Lesion Substudy: Long Lesions Substudy Cohort will evaluate the safety and effectiveness of the ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.
- PK Substudy: PK Substudy Cohort will evaluate the safety and pharmacokinetics of the ELUVIA stent for the treatment of atherosclerotic lesion(s) up to 140 mm in length in the SFA/PPAPK. Time-points for analysis are baseline venous blood drawn followed by blood draws at 10 minutes, 30 minutes, 1, 2, 3, 4, 6, 12, and 24 hours and one final blood draw at either 48 hours or 72 hours after placement of the ELUVIA stent.
Period: Overall Study
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Started | 309 | 156 | 50 | 13
Completed | 195 | 102 | 25 | 8
Not Completed | 114 | 54 | 25 | 5
Not completed — Withdrawal by Subject | 29 | 15 | 4 | 1
Not completed — Adverse Event | 5 | 1 | 1 | 0
Not completed — Visit Missed | 15 | 7 | 5 | 0
Not completed — Other | 7 | 2 | 0 | 0
Not completed — Death | 48 | 26 | 12 | 4
Not completed — Physician Decision | 5 | 2 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Long Lesion Substudy: Long Lesion Substudy Cohort will evaluate the safety and effectiveness of the ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.
- Total: Total of all reporting groups
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy | Total
Number analyzed (Participants) | 309 | 156 | 50 | 13 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (9.5) | 67.8 (9.4) | 68.2 (8.9) | 66.4 (6.1) | 68.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 52 | 18 | 3 | 178
  Male | 204 | 104 | 32 | 10 | 350
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 6 | 3 | 0 | 27
  Caucasian | 205 | 108 | 30 | 13 | 356
  Asian | 1 | 0 | 0 | 0 | 1
  Japanese | 56 | 28 | 11 | 0 | 95
  Black, or African Heritage | 21 | 11 | 6 | 0 | 38
  Native Hawaiian or Pacific Islander | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 2 | 2 | 0 | 0 | 4
  Other | 3 | 1 | 0 | 0 | 4
  Not Disclosed | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  New Zealand | 9 | 5 | 1 | 0 | 15
  Canada | 17 | 7 | 0 | 0 | 24
  Europe | 89 | 44 | 4 | 0 | 137
  United States | 138 | 72 | 34 | 13 | 257
  Japan | 56 | 28 | 11 | 0 | 95
History of Smoking (Current) [Count of Participants; unit: Participants] | 109 | 63 | 16 | 3 | 191
History of Smoking (Previous) [Count of Participants; unit: Participants] | 157 | 68 | 26 | 10 | 261
History of Smoking (Never) [Count of Participants; unit: Participants] | 42 | 22 | 8 | 0 | 72
History of Smoking (Unknown) [Count of Participants; unit: Participants] | 1 | 3 | 0 | 0 | 4
Current Diabetes Mellitus [Count of Participants; unit: Participants] | 129 | 68 | 20 | 7 | 224
History of Hyperlipidemia requiring medication [Count of Participants; unit: Participants] | 235 | 118 | 41 | 12 | 406
History of Hypertension requiring medication [Count of Participants; unit: Participants] | 254 | 133 | 46 | 12 | 445
History of Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] | 48 | 28 | 9 | 2 | 87
History of Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 156 | 70 | 28 | 7 | 261
History of Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 60 | 27 | 9 | 2 | 98
History of Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 26 | 12 | 8 | 1 | 47
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 100 | 53 | 18 | 3 | 174
History of Coronary Artery Bypass Surgery (CABG) [Count of Participants; unit: Participants] | 43 | 21 | 7 | 3 | 74
Stable Angina [Count of Participants; unit: Participants] | 32 | 19 | 5 | 0 | 56
History of Transient Ischemic Attacks (TIA) [Count of Participants; unit: Participants] | 14 | 6 | 5 | 1 | 26
History of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] | 30 | 14 | 9 | 4 | 57
History of Renal insufficiency [Count of Participants; unit: Participants] | 25 | 11 | 3 | 2 | 41
History of Renal Percutaneous Intervention [Count of Participants; unit: Participants] | 6 | 1 | 0 | 0 | 7
History of Peripheral Vascular Surgery [Count of Participants; unit: Participants] | 40 | 15 | 2 | 1 | 58
History of endovascular interventions in Target Vessel [Count of Participants; unit: Participants] | 27 | 17 | 2 | 1 | 47
History of Other Peripheral Endovascular Interventions (other than Target Vessel) [Count of Participants; unit: Participants] | 112 | 49 | 20 | 5 | 186
History of Claudication [Count of Participants; unit: Participants] | 303 | 151 | 49 | 13 | 516

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Adverse Events (MAEs)
Description: MAEs defined as all causes of death through 1 month, target limb major amputation through 12 months and/or target lesion revascularization (TLR) through 12 months
Time Frame: 12 Months
Measure: Number; unit: percentage of participants
Groups:
- Long Lesion Substudy: To evaluate the safety and effectiveness of the Boston Scientific Corporation (BSC) ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.
- PK Substudy: To further evaluate the safety and pharmacokinetics of the ELUVIA stent for the treatment of atherosclerotic lesion(s) up to 140 mm in length in the SFA/PPAPK. Time-points for analysis are baseline venous blood drawn followed by blood draws at 10 minutes, 30 minutes, 1, 2, 3, 4, 6, 12, and 24 hours and one final blood draw at either 48 hours or 72 hours after placement of the ELUVIA stent.
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 287 | 132 | 50 | 13
percentage of participants
  All Causes of Death at 1 Month | 0 | 0 | 0 | 0
  Target Limb Major Amputation | 0.3 | 0 | 0 | 0
  Target Lesion Revascularization | 4.5 | 9.0 | 6.5 | 0
Statistical Analysis 1: Comparison: ELUVIA Stent Implantation vs Zilver PTX Stent Implantation; Test type: Non-Inferiority — A two-group Farrington-Manning test is used to test the one-sided hypothesis of non-inferiority in proportions; p < 0.0001, Farrington-Manning — A two-group Farrington-Manning test is used to test the one-sided hypothesis of non-inferiority in proportions. If the P-value from the one-sided Farrington-Manning test is <0.05, Eluvia is concluded to be non-inferior to Zilver PTX

2. Primary Outcome: Number of Participants Reaching Primary Patency
Description: Primary patency of target lesion at 12-months assessed by duplex ultrasound and adjudicated by an independent core laboratory
Time Frame: 12 Months
Population: Primary Patency: percentage (%) of lesions (target stented segments) that reach endpoint without a hemodynamically significant stenosis on DUS and without clinically-driven TLR or, bypass of the target lesion before or on the DUS FU visit. Per PK sub-study design, primary efficacy (patency) not analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Long Lesion Substudy: To evaluate the safety and effectiveness of the ELUVIA Drug-Eluting Vascular Stent System (ELUVIA Stent) for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.
- PK Substudy: To evaluate the safety and pharmacokinetics of the ELUVIA stent for the treatment of atherosclerotic lesion(s) up to 140 mm in length in the SFA/PPAPK. Time-points for analysis are baseline venous blood drawn followed by blood draws at 10 minutes, 30 minutes, 1, 2, 3, 4, 6, 12, and 24 hours and one final blood draw at either 48 hours or 72 hours after placement of the ELUVIA stent.
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 266 | 130 | 46 | 0
Participants | 231 | 106 | 40 |
Statistical Analysis 1: Comparison: ELUVIA Stent Implantation vs Zilver PTX Stent Implantation; Test type: Non-Inferiority — A two-group Farrington-Manning test is used to test the one-sided hypothesis of non-inferiority in proportions; p < 0.0001, Farrington-Manning — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of CEC-adjudicated Events Through 12 Months
Description: Denominators for the cumulative rate will be based on 1) subjects with events, and 2) subjects with no events but their follow-up time reach on (or beyond) the earliest visit window.
Time Frame: 12 Months
Population: Denominators for the cumulative rate will be based on 1) subjects with events, and 2) subjects with no events but their follow-up time reach on (or beyond) the earliest visit window.
Measure: Number; unit: participants
Groups:
- Long Lesion Substudy: To evaluate the safety and effectiveness of the ELUVIA Stent for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions >140 mm and ≤ 190 mm in length.
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 292 | 150 | 46 | 13
participants
  All deaths | 6 | 6 | 0 | 0
  Target Lesion Revascularization | 13 | 13 | 3 | 1
  Target Vessel Revascularization | 20 | 13 | 4 | 0
  Target Limb Amputation | 1 | 2 | 0 | 0
  Stent Thrombosis | 5 | 6 | 0 | 0

4. Secondary Outcome: Count of Participants Meeting Primary Sustained Clinical Improvement
Description: Defined as improvement in Rutherford classification (defined as chronic, symptomatic lower limb ischemia in categories 2, 3 or 4) by one or more categories compared with baseline, without target lesion revascularization.
Time Frame: 12 Months
Population: Per PK sub-study design, secondary endpoint not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 279 | 142 | 47 | 0
Participants | 250 | 118 | 35 |

5. Secondary Outcome: Number of Participants With Hemodynamic Improvement
Description: Defined as an increase in the ankle-brachial index by greater than of equal to 0.10 compared with baseline or to an ankle-brachial index of greater than or equal to 0.90, without need for repeat target lesion revascularization.
Time Frame: 12 Months
Population: Per PK sub-study design, secondary endpoint not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 276 | 141 | 45 | 0
Participants | 223 | 111 | 37 |

6. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Scores
Description: The WIQ is a functional-assessment questionnaire that evaluates walking ability with regard to speed, distance and stair climbing ability as well as the reasons that walking ability might be limited. Range of scores is between 0% and 100% with 100% being the best and 0% being the worst score. WIQ scores reported as change from baseline.
Time Frame: Baseline to 12 Months
Population: Not all subjects were able to complete questionnaires.Per PK sub-study design, secondary endpoint not analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 279 | 141 | 47 | 0
Units on a scale
  Distance | 33.16 (38.33) | 29.49 (38.19) | 58.67 (36.60) |
  Speed: number analyzed (Participants) | 277 | 141 | 47 | 0
  Speed | 18.25 (29.46) | 18.08 (28.72) | 41.21 (25.95) |
  Stair climbing: number analyzed (Participants) | 276 | 140 | 47 | 0
  Stair climbing | 19.43 (36.68) | 21.10 (34.55) | 56.29 (34.55) |

7. Secondary Outcome: 6-Minute Walk Test - Distance Walked
Description: Change in distance walked from baseline to 12 months.
Time Frame: Change in baseline to 12-Months
Population: Per PK sub-study design, secondary endpoint not analyzed.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 269 | 136 | 42 | 0
m | 323.8 (148.5) | 323.4 (155.4) | 293.5 (123.8) |

8. Secondary Outcome: 6-Minute Walk Test - Speed
Description: Change in speed walked from baseline to 12 months
Time Frame: Baseline to 12 months
Population: Per PK sub-study design, secondary endpoint not analyzed.
Measure: Mean (Standard Deviation); unit: m/min
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 269 | 136 | 42 | 0
m/min | 55.5 (23.3) | 56.1 (24.1) | 50.3 (19.3) |

9. Other Pre Specified Outcome: Freedom From Major Adverse Events
Description: Percentage of participants without Major Adverse Events (MAEs)
Time Frame: Through 60 Months
Population: PK Substudy cohort was not included in this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 232 | 114 | 35 | 0
Participants | 156 | 74 | 19 | 0

10. Other Pre Specified Outcome: Clinical Events Committee Adjudicated Clinically-Driven Target Lesion Revascularization Rate
Description: Clinical Events Committee (CEC) adjudicated clinically-driven target lesion revascularization rate
Time Frame: Through 60 Months
Population: PK Substudy cohort was not included in this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 273 | 139 | 46 | 0
Participants | 68 | 39 | 15 | 0

11. Other Pre Specified Outcome: Percentage of Participants With Target Limb Major Amputation
Description: Clinical Events Committee (CEC) adjudicated target limb major amputation rate
Time Frame: Through 60 Months
Population: PK Substudy cohort was not included in this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
Number analyzed (Participants) | 273 | 139 | 46 | 0
Participants | 8 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected to five year (60M) post-implant.
Arm/Group | ELUVIA Stent Implantation | Zilver PTX Stent Implantation | Long Lesion Substudy | PK Substudy
All-Cause Mortality (participants affected / at risk) | 58/309 | 28/156 | 13/50 | 6/13
Serious Adverse Events (participants affected / at risk) | 243/309 | 126/156 | 40/50 | 13/13
Other Adverse Events (participants affected / at risk) | 186/309 | 91/156 | 27/50 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELUVIA Stent Implantation (N=309) | Zilver PTX Stent Implantation (N=156) | Long Lesion Substudy (N=50) | PK Substudy (N=13)
Peripheral artery stenosis (Vascular disorders) | 85 (144) | 42 (73) | 10 (14) | 2 (2)
Intermittent claudication (Vascular disorders) | 36 (55) | 13 (20) | 9 (14) | 2 (9)
Peripheral arterial occlusive disease (Vascular disorders) | 27 (42) | 15 (19) | 3 (4) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 27 (35) | 6 (8) | 4 (4) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 14 (19) | 4 (4) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 3 (3) | 2 (3) | 1 (1) | 1 (2)
Haematoma (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 5 (7) | 8 (9) | 2 (2) | 1 (1)
Aortic aneurysm (Vascular disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 14 (18) | 8 (9) | 2 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 15 (16) | 4 (4) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 16 (17) | 6 (6) | 1 (1) | 1 (1)
Cardiac Failure (Cardiac disorders) | 14 (15) | 5 (5) | 5 (6) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 13 (15) | 6 (6) | 2 (2) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 4 (5) | 3 (4) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 6 (11) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (9) | 3 (3) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 6 (7) | 1 (1) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tricuspid valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 16 (19) | 15 (17) | 8 (10) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 4 (6) | 2 (5) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 5 (6) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 3 (4)
Urosepsis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (7) | 0 (0) | 0 (0)
Intervetebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5) | 1 (1) | 2 (4) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 7 (7) | 5 (5) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 7 (9) | 2 (2) | 2 (2) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 6 (7) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 3 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (3) | 0 (0) | 2 (2) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 9 (9) | 4 (4) | 2 (2) | 1 (1)
Chest pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 4 (6) | 0 (0) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Therapeutic response decreased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Treatment failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 10 (12) | 2 (3) | 1 (1) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
B-Cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (3) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 7 (8) | 4 (4) | 0 (0) | 2 (2)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoperfusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Invertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (5) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvar dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulse absent (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial septal defect acquired (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Listeria sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELUVIA Stent Implantation (N=309) | Zilver PTX Stent Implantation (N=156) | Long Lesion Substudy (N=50) | PK Substudy (N=13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (13) | 6 (7) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 2 (2) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 18 (22) | 6 (6) | 3 (3) | 0 (0)
Intermittent claudication (Vascular disorders) | 10 (10) | 11 (11) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 5 (5) | 2 (2) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6) | 3 (3) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arterial spasm (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 16 (16) | 9 (10) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 12 (12) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (8) | 2 (4) | 0 (0) | 1 (1)
Chest pain (General disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disuse syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (5) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebellar atrophy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periventricular leukomalacia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudoradicular syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculitis cerival (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 8 (8) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presbyacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal bruit (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint prosthesis user (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tarsi syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle brachial index decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infected bunion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02574481/Prot_SAP_000.pdf